CLINICAL TRIAL: NCT06397859
Title: Effectiveness and Clinical Outcomes of Long-term Bulevirtide Monotherapy in Patients With HDV-related Compensated Cirrhosis (SAVE-D Study)
Brief Title: Effectiveness and Clinical Outcomes of Long-term Bulevirtide Monotherapy in Patients With HDV-related Compensated Cirrhosis
Acronym: SAVE-D
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: IN-IT-589-7118
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-04

CONDITIONS: Hepatitis D
MeSH Terms: conditions — Hepatitis D | interventions — bulevirtide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hepatis Delta: Bulevirtide (BLV) at a dose of 2 mg/day subcutaneously
  Interventions: Drug: Bulevirtide

INTERVENTIONS:
Drug: Bulevirtide — dose of 2 mg/day subcutaneously
  Other Names: Hepcludex

SUMMARY:
Retrospective and prospective, pharmacological, multicentre, non-profit observational study.

Consecutive patients with HDV-related compensated cirrhosis starting Bulevirtide 2 mg/day from September 2019 to December 2025 will be enrolled in the study.

Aim of this study is to investigate virological and clinical effectiveness of Bulevirtide 2 mg/day in patients with HDV-related compensated cirrhosis in the real-life setting.

Primary endpoint of the study is the rate of virological response, defined as at least 2 Log decline or undetectable HDV RNA compared to baseline, at week 96 of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years
* HDV-related compensated cirrhosis defined by positivity of HDV RNA for at least 6 months and clinical or laboratory or histological diagnosis of cirrhosis
* Started treatment with BLV monotherapy between September 1st 2019 and 2025

Exclusion Criteria:

* Chronic hepatitis without any evidence of cirrhosis
* Decompensated cirrhosis
* PegIFN alpha therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enrol patients with chronic HDV infection (defined by HDV RNA positivity for at least 6 months) who started or will start BLV 2 mg/day during the study period at the S.C. Gastroenterology and Hepatology (Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico) and at participating centers, and who meet the inclusion criteria and do not present any of the exclusion criteria. The decision to treat patients with BLV is determined based on the clinical judgment of the treating physicians prior to study enrolment.
Sampling Method: Non-Probability Sample
Enrollment: 266 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Investigate the virological response rate to BLV | Week 96
  Percentage of patients with >2 Log decline in HDV-RNA (IU/mL)
Investigate the virological response rate to BLV | Week 96
  Percentage of patients with undetectable HDV-RNA (IU/mL)

SECONDARY OUTCOMES:
Evaluation of the proportion of patients with virological response, defined as a >2 Log decline in HDV-RNA (IU/mL) or undetectable HDV-RNA (IU/mL) along with normalization of ALT (combined response) | Week 96
  Percentage of patients with >2 Log decrease in HDV-RNA along with normalization of ALT (combined response)
Evaluation of the percentage of patients with normal ALT | Week 96
  Percentage of patients with normal ALT
Evaluation of the percentage of patients with <1 Log decrease in HDV-RNA | Week 96
  Percentage of patients with < 1 log decline HDV RNA levels
Evaluation of the percentage of patients with clinical response, i.e., the percentage of patients who remain free of liver complications, such as HCC or decompensation, at week 96 of treatment. | Week 96
  Percentage of patients who remain free of liver complications (de novo HCC or onset of decompensation) at week 96;
Evaluation of the correlation between baseline or on-treatment biochemical/clinical variables and virological response | Week 96
  Baseline and on-treatment biochemical and clinical variables predicting virological response to BLV
Evaluation of virological and clinical responses from year 2 (week 96) to year 5 only (only if data of this patients is available) | Year 5
  Percentage of patients with virological, biochemical and clinical responses from year 2 (week 96) to year 5
Evaluation of bile acids levels over time and correlation of bile levels with virological response rates | Week 96
  Correlation between bile acids levels and virological response over time

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation IRCCS Ca' Granda Ospedale Maggiore Policlinico, Division of Gastroenterology and Hepatology, Milan, Italy., Milan, Italy